CLINICAL TRIAL: NCT00214266
Title: A Pilot Study of Campath-1H Induction Therapy Combined With CellCept® Therapy to Allow for a Calcineurin Inhibitor Free Regimen After Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2004-0209
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Alemtuzumab; Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Campath-1H Induction Therapy Combined With CellCept® Therapy (Experimental): Campath-1H Induction Therapy Combined With CellCept® Therapy
  Interventions: Drug: Campath 1H®, Rituximab, mycophenolate mofetil

INTERVENTIONS:
Drug: Campath 1H®, Rituximab, mycophenolate mofetil — Induction therapy with Campath 30mg IV x 2 doses, Rituximab 375mg/m2 x 1, corticosteroids, and mycophenolate 1000mg bid

SUMMARY:
The hypothesis of this study is that lymphocyte depletion by Campath-1H and rituximab will obviate the need for long-term calcineurin inhibitors in renal transplantation. Most successful strategies to date have relied on the use of either tacrolimus or cyclosporine. However, the advantage of a calcineurin inhibitor free regimen may include improved renal allograft function, a lower incidence of hypertension, diabetes, and less drug related side effects. This is a non-randomized open-label pilot trial in 30 adult renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipients

Exclusion Criteria:

* Recipients of HLA-identical living-donor renal transplants;
* multi-organ transplant;
* known hypersensitivity to Campath-1H, Rituximab, CellCept, or prednisone;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
renal allograft function | 2 years

SECONDARY OUTCOMES:
incidence of hypertension | 2 years
incidence of diabetes | 2 years
drug related side effects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Sollinger, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States